CLINICAL TRIAL: NCT01470183
Title: Lupus Nephritis Biomarker Study: Baseline Characteristics of Patients
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Centocor Research & Development, Inc. (Industry)
Responsible Party: Principal Investigator, Gerald B. Appel, Professor of Clinical Medicine, Nephrology, Columbia University
Other Study IDs: AAAI1090
Record Dates: First submitted 2011-11-07; First posted 2011-11-11 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lupus Nephritis Patients: 1. Male or female subjects age 18 and older
  2. Must have confirmed diagnosis of Class III or Class IV lupus nephritis by biopsy
  3. Must have stable disease on medication at time of enrollment
- Control Patients: Any patient with an idiopathic glomerular disease who does not have lupus nephritis. This includes patients with minimal change disease, membranous nephropathy, focal segmental glomerulosclerosis, and IgA nephropathy.

SUMMARY:
This is an exploratory study. No formal hypothesis will be tested.

The objectives of this study are to follow Lupus Nephritis patients over a period of 12 months to:

* Establish the baseline biomarker characteristics of patients
* Determine the variability of biomarker measures over time
* Correlate biomarkers with disease phenotype

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 80 years of age, inclusive
* Diagnosis of SLE by ACR criteria and biopsy-proven ISN/RPS Class III or IV lupus glomerulonephritis within 2 years
* Persistently active nephritis defined as proteinuria greater than or equal to 1.0 g/day for 3 months or more, AND at least 1 of the following:

  * Hematuria (greater than or equal to 5 RBC/hpf) on 2 or more urinalyses done greater than or equal to 2 weeks apart
  * anti-dsDNA positive or anti-Smith positive, or
  * low C3 or C4 complement level. (d) Stable immunosuppression consisting of mycophenolate mofetil (MMF) 13 g/day with/without corticosteroids up to prednisone equivalent of 15 mg/day, or azathioprine 13 mg/kg/day with/without corticosteroids up to prednisone equivalent of 20 mg/day.
* Stable dose of ACE inhibitor/ARB for 4 weeks prior to study enrollment, unless previously intolerant to or having a contraindication to ACE inhibitors and ARBs
* If using oral corticosteroids, must be on a stable dose equivalent to less than or equal to 15 mg/day of prednisone for at least 4 weeks prior to study enrollment. If currently not using corticosteroids, the subject must not have received oral corticosteroids for at least 4 weeks prior study enrollment.
* Clarification of inclusion criteria for controls: Any patient with an idiopathic glomerular disease who does not have lupus nephritis. This includes patients with minimal change disease, membranous nephropathy, focal segmental glomerulosclerosis, and IgA nephropathy.

Exclusion Criteria:

* B-cell depletion therapy in past 1 yr, or evidence of persistent B cell depletion at the time of screening.
* Received an investigational drug (including vaccines) or used an investigational medical device within 3 months of study enrollment or within 5 half-lives of agent, whichever is longer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 50 adult patients, 25 with lupus nephritis 25 control patients who have greater than 1 gram per day proteinuria and non-SLE diagnoses, and who qualify for this study based upon the stated inclusion/exclusion criteria will be recruited from the Glomerular Center at Columbia University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in mRNA | Week 0, and Months 1, 2, 4, 6, 8, 10 and 12
  Whole blood samples will be collected from all subjects for the analysis of mRNA expression of genes relevant to lupus nephritis (IFNa signature, TNFa/TNFa receptor families, defensins, TH1, TH17 related pathway genes.
Change in Proteinuria | Week 0, and Months 1, 2, 4, 6, 8, 10 and 12
  Urine (12-hour collections) will be obtained from all subjects in the study for the analysis of proteins relevant to lupus nephritis.
Change in Creatinine | Week 0, and Months 1, 2, 4, 6, 8, 10 and 12
  Serum will be collected from all subjects in the study for the analysis of proteins relevant to lupus nephritis.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Appel, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, Division of Nephrology, Glomerular Center, New York, New York, United States